CLINICAL TRIAL: NCT03121560
Title: Acceptability and Tolerance of Hysteroscopy and Hysterosonography in Consultation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Andre Nazac, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-EVAdolHYSIS
Record Dates: First submitted 2017-04-14; First posted 2017-04-20 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Metrorrhagia
Keywords: Hysteroscopy; Saline infusion hysterosonography
MeSH Terms: conditions — Metrorrhagia | interventions — Hysteroscopy

STUDY DESIGN:
Intervention Model Description: Prospective cross-over study (each woman will be her own control) on women with peri-menopausal menorrhagia. Each woman, after signing the informed consent, will come into the "bleeding clinic" where she will undergo both examinations in a random order, in two days time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hysteroscopy (Active Comparator): Women with ≥ 18 with abnormal bleeding (post-menopausal menorrhagia or metrorrhagia), managed at bleeding clinic. Each women will undergo an hysteroscopy and a hysterosonography and will be her own control.
  Interventions: Device: Hysteroscopy
- Hysterosonography (Experimental): Women with ≥ 18 with abnormal bleeding (post-menopausal menorrhagia or metrorrhagia), managed at bleeding clinic. Each women will undergo an hysteroscopy and a hysterosonography and will be her own control.
  Interventions: Device: Hysterosonography

INTERVENTIONS:
Device: Hysteroscopy — Hysteroscopy allows a direct visualization of the interior of the uterine cavity in order to invalidate or confirm the presence of uterine pathologies.In the pre-menopausal period, it is preferable to perform a hysteroscopy at the beginning of the follicular phase (just after the menstruations, when the endometrium is atrophic). Use of a rigid hysteroscope comprising a 2.9 mm optics and a 4.3 mm sheath with a 5 - bit operator channel allowing the realization of a biopsy.
  Arms: Hysteroscopy
Device: Hysterosonography — Hysterosonography (SIS) is an endovaginal ultrasound performed along with an injection of saline in order to observe the uterine cavity and detect any endometrial pathology. A 3D image can be associated with it to define the topography of a lesion. It is ideally performed in the first part of the cycle. Use of the GE Voluson E8 Ultrasound System.
  Arms: Hysterosonography

SUMMARY:
Menorrhagia is frequent and occur in 11 to 13 % of the general population. It accounts for 20% of the gynecological consultations and tends to increase with age. It can be the first symptom of a mild uterine disease or cancer (cervical or endometrial), especially if the patient is older. The most common causes are polyps, adenomyosis, fibroids, hyperplasia and cancer.

Menorrhagia needs to be investigated -especially after menopause, when the prevalence of endometrial cancer is higher (10-15%). For premenopausal metrorrhagia, the assessment will be made if a pathology is suspected or if there is no response to the medical treatment within 3 to 6 months.

The medical check-up consists in the first instance in a questionnaire, a clinical examination and an endovaginal ultrasound examination. If the endometrium is thickened, a focal pathology is suspected, or if the bleeding persists despite a normal endovaginal ultrasound result, further examinations including a possible biopsy are required.

While hysteroscopy is widely accepted as a standard examination for uterine cavity exploration, a meta-analysis showed that the diagnostic performance of hysterosonography was equivalent. Both are carried out on an outpatient basis during a gynecological consultation and require no special preparation. Several studies seem to show that hysterosonography is less painful, causes less discomfort and is therefore more accepted by patients than hysteroscopy. This is why many practitioners continue to prefer it to hysteroscopy and associate it with the Pipelle of Cornier for the assessment of postmenopausal metrorrhagia.

However, if endometrial cancer is confirmed, the histological type detected within the biopsy is the main predictor of the severity of the disease and the treatment to be given. It is therefore essential to have an accurate biopsy sampling prior to therapeutic management. It is not the case with blind biopsies (without visual control). Indeed, some studies showed that the concordance between the optical aspect of the endometrium under hysteroscopy and the histological result was close to 90%, validating the hypothesis of an improved sensitivity through visual control.

The American College of Obstetricians and Gynecologists (ACOG) currently recommends an endovaginal ultrasound assessment followed by an endometrial biopsy in the event of a thickened endometrium or when a pathology is suspected. A biopsy can even be taken during the consultation, at the onset of the complaints. The last recommendations of December 2010 leave the choice to clinicians regarding the histological diagnostic modalities (a blind biopsy with the Pipelle of Cornier or a targeted biopsy under hysteroscopy), although the biopsies under hysteroscopy are recommended since 2015. However, despite its poor sensitivity, the most widely used technique in the world is the blind biopsy by aspiration performed after vaginal ultrasound or hysterosonography because it is an easy low cost method.

The development of hysteroscopes with a smaller diameter and the introduction of the vaginoscopy have considerably increased the tolerance of this examination. In addition, hysteroscopy allows a simultaneous therapeutic intervention for certain indications, which is comfortable and well accepted by the patients. Unfortunately, there are few studies comparing the tolerance of the two examinations performed according to the current recommendations of good practice of hysteroscopy. Only one comparative randomized study in 2008 showed that saline infusion sonography (SIS) was less painful than hysteroscopy with vaginoscopy. However, direct comparison was impossible since women only had one of the two examinations.

The Brugmann University Hospital set up a consultation called "one stop bleeding clinic" in which the two examinations are performed for each patient with abnormal bleedings, in order to increase diagnostic performance.

All included patients will thus undergo a saline infusion sonography (SIS) and a hysteroscopy (HSC). Each procedure will be evaluated on pain level (EVA scale) and tolerance by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Women with abnormal bleedings (post-menopausal menorrhagia or metrorrhagia managed at bleeding clinic) without endometrial measurement criteria.
* Level of French/Dutch sufficient to understand the informed consent document and the pain evaluation scale

Exclusion Criteria:

* Spontaneous intake of an analgesic before the examinations
* Women who already had an SIS or hysteroscopy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
EVA pain scale | Baseline: before the examination
  Visual analogic pain scale. It is a graduated horizontal or vertical scale of 10 cm with 2 marks: 0 for the complete absence of pain and 10 for the worst lived pain.
EVA pain scale | 1 minute after the examination
  Visual analogic pain scale. It is a graduated horizontal or vertical scale of 10 cm with 2 marks: 0 for the complete absence of pain and 10 for the worst lived pain.
EVA pain scale | 5 minutes after the examination
  Visual analogic pain scale. It is a graduated horizontal or vertical scale of 10 cm with 2 marks: 0 for the complete absence of pain and 10 for the worst lived pain.

SECONDARY OUTCOMES:
Number of side effects | 2 days
  Number of side effects for each technique
Patient tolerance | 2 days
  Patients will be asked at the end of the consultation if they would be ready to repeat the experiment or if they would have preferred to have the examination under general anesthesia.
Histological diagnose performance of each technique | 2 days
  Histological diagnostic performance (sensitivity and specificity) of each technique (biopsies)
Examination duration | 2 days
  Comparison of the duration of the two techniques

CONTACTS AND LOCATIONS:
Overall Officials: André Nazac, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No